CLINICAL TRIAL: NCT04668118
Title: The Effect of 3% Diquafosol Ophthalmic Solution on Visual Display Terminal-associated Dry Eye
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Diquafosol
Record Dates: First submitted 2020-12-06; First posted 2020-12-16 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-04

CONDITIONS: Dry Eye Syndromes; Computer Vision Syndrome; Asthenopia
MeSH Terms: conditions — Dry Eye Syndromes; Asthenopia | interventions — diquafosol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diquafosol group (Experimental): The treatment period is 12 weeks. The day after subjects who meet the inclusion criteria undergo baseline examination is the day starting the medication. Dosing frequency was six times daily for 3% Diquafosol Ophthalmic Solution. The follow-up time points are 2, 4, 8, 12 weeks, and no other medication is required on the follow-up day.
  Interventions: Drug: Diquafosol

INTERVENTIONS:
Drug: Diquafosol — As a P2Y2 receptor agonist, diquafosol can be used to stabilize the tear film by stimulating P2Y2 receptors on the corneal epithelial cells and conjunctival goblet cell, which increase the secretion of tear fluid and mucin on the ocular surface, thereby repairing the ocular surface and stabilizing the tear film.
  Other Names: Diquafosol Sodium Eye Drops; 3% Diquafosol Ophthalmic Solution

SUMMARY:
This study aims to evaluate the efficacy and safety of 3% Diquafosol Ophthalmic Solution for visual display terminal (VDT)-associated dry eye and to investigate the mechanism of treatment.

DETAILED DESCRIPTION:
The treatment period is 12 weeks. The day after subjects who meet the inclusion criteria undergo baseline examination is the day starting the medication. The dosing frequency was six times daily for 3% Diquafosol Ophthalmic Solution. The follow-up time points are 2, 4, 8, 12 weeks, and the investigator will evaluate the symptoms and signs of Dry Eye.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with a diagnosis dry eye based on Chinese Dry Eye Diagnosis Standard (2020)；
* Working in the offices with VDTs more than 4h daily；
* Working in the offices with VDTs at least five days per week；
* Provision of written informed consent.

Exclusion Criteria:

* Known allergy to any eye drops
* Ocular therapies other than artificial tears
* Presence of any of the following conditions: active ocular infection, ocular inflammation, active ocular allergy, contact lens wear, ocular surgical history, laser treatment in the last 3 months, Meibomian gland dysfunction (MGD) over grade 2 (the grade is according to the report of the International Workshop on MGD in 2011), severe blepharitis or obvious inflammation of the eyelid margin, which in the judgment of the investigator may interfere with the interpretation of the study results
* Pregnant and lactating women, or those planning a pregnancy over the course of the study
* Uncontrolled systemic disease
* Hypersensitivity or intolerance to diquafosol(DQS)
* Subjects with a history of anxiety and depression

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-03-25 (Estimated)

PRIMARY OUTCOMES:
the changes of Ocular Surface Disease Index (OSDI) scores | 12 weeks after intervention
  OSDI is one of the most frequently used questionnaires for evaluation of Dry eye disease(DED). This includes 12 questions which measure the frequency of symptoms over the recent week, and the scores range from 0 to 100. The higher the score, the worse the result.
the changes of Tear break-up time (TBUT) | 12 weeks after intervention
  TBUT is the time from normal blinking to the first appearance of a break in the tear film. The BUT was measured using fluorescein with a metronome, and the average of three consecutive BUTs was calculated. The shorter the TBUT, the worse the outcome.

SECONDARY OUTCOMES:
the changes of scores of Corneal fluorescein staining (CFS) | 12 weeks after intervention
  The degree of fluorescein staining of the cornea was evaluated using the National Eye Institute (NEI) scale of five corneal regions (central, superior, temporal, nasal, and inferior). The degree of staining in each of the five regions was graded on a scale of 0-3 according to the NEI/Industry Workshop method: 0 =no staining, 1 =mild staining, 2 = moderate staining, and 3 = severe staining. The maximal score for each area was 3. The scores of the five areas were added to obtain a total score for each eye. The higher the score, the worse the result.
the changes of scores of Lissamine green staining | 12 weeks after intervention
  To grade the temporal zone, the subject looks nasally; to grade the nasal zone the subject looks temporally. The upper and lower conjunctiva can also be graded. The higher the score, the worse the result.
the changes of value of Schirmer Ⅰ test (SⅠt) | 12 weeks after intervention
  The Schirmer I test is performed using sterile strips without anesthesia. The strips are placed in the lateral part of the inferior fornix of the eye for 5min and the extent of tear flow down was measured in millimeters. The higher the value, the better the result.
the changes of Lipid layer thickness(LLT) | 12 weeks after intervention
  Lipid layer is evaluated by Lipiview interferometer (TearScience Inc, Morrisville, NC, USA) which records a 15-s live digital image of the interference pattern of the tear film. The interferometry color units (ICU) of the tear film which is an indicator of lipid layer thickness is assessed according to the mean interference color pattern through specular reflection. The higher the thickness, the better the result.
the changes of Partial blink rate(PBR) | 12 weeks after intervention
  PBR can be provided by Lipiview interferometer, which mainly evaluate incomplete blinking. The higher the rate, the worse the result.

CONTACTS AND LOCATIONS:
Overall Officials: Tingting Yang, MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China